CLINICAL TRIAL: NCT02926547
Title: New Approaches for the Identification and Characterization of Functional Markers of the Risk of Extension of Breast Cancer Without Lymph Node Involvement
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2011/PR-01
Record Dates: First submitted 2016-09-09; First posted 2016-10-06 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: proteomics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — This proteomic study is performed on biological samples originally as part of a diagnostic approach reclassified in the absence of opposition from patients, from the Biobank of Nîmes University hospital (Ministry of Higher Education and Research No. AC-2008-107; South Mediterranean CPP III No. COL2008.04.02).
  For validation part, the investigators will work on sections of TMA already made from samples drawn between 2000 and 2003.

GROUPS / COHORTS (2):
- CCIS
- invasive breast cancer

SUMMARY:
1. Identify the tissue proteins associated with early breast cancer invasion phases without lymph node involvement .
2. Consider their role in the invasion and the risk of tumor spread .

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* CCIS
* Invasive tumors
* Breast cancer tissues available in the biobank

Exclusion Criteria:

* non availability of cancer tissue specimen

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CCIS and invasive breats cancer in women
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
A list of the ten proteins most associated with early breast cancer invasion phases without lymph node involvement . | Day 0
  The primary objective of this study is to Identify the tissue proteins associated with early breast cancer invasion phases without lymph node involvement. The outcome is a list of identified proteins.